CLINICAL TRIAL: NCT04854811
Title: A Proof of Concept Phase II Study With the PDE4 Inhibitor Roflumilast in People Suffering From Long-term Cognitive Sequela After Stroke
Brief Title: Roflumilast to Treat Cognitive Sequela After Stroke
Acronym: ROSTMEMA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Maastricht University (Other)
Collaborators: Netherlands Brain Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NL74897.068.20
Record Dates: First submitted 2021-03-31; First posted 2021-04-22 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Cerebrovascular Disorders; Memory; Functional Recovery; Drug Intervention
Keywords: Cerebrovascular Disorders; Plasticity; Phosphodiesterase inhibitor; Memory; Roflumilast
MeSH Terms: conditions — Cerebrovascular Disorders | interventions — Roflumilast; Phosphodiesterase 4 Inhibitors

STUDY DESIGN:
Intervention Model Description: Between subjects, double blind, placebo-controlled, randomized
Who Masked: Participant, Investigator
Masking Description: Pharmacy will distribute pills with a code
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo oral capsule, once daily for 12 weeks
  Interventions: Drug: Roflumilast Oral Tablet
- Roflumilast (100 microgram) (Experimental): once daily for 12 weeks
  Interventions: Drug: Roflumilast Oral Tablet

INTERVENTIONS:
Drug: Roflumilast Oral Tablet — Once daily for 12 weeks
  Other Names: EU: Daxas; US: Daliresp; PDE4 inhibitor

SUMMARY:
The aim of the current project is to validate the effects of chronic rolflumilast treatment (12 weeks) on cognitive functions (i.e. episodic memory) by means of behavioral tasks, in people suffering from cognitive impairments at least 1 year after stroke. Secondarily, the effects of roflumilast on daily activities and well-being will be assessed.

DETAILED DESCRIPTION:
Rationale: In the Netherlands there are about 400.000 people who suffer from long-term consequences of a stroke. In the first months, spontaneous neurological recovery can take place, but there is hardly any functional recovery found one year after a stroke. About 40% of these patients indicate that one of the greatest problems they are facing is the impairment in cognitive functions, which also seems to be predictive for the disease outcome. Currently, the main focus of helping these patients is helping them to cope with and adapt to the new situation. There is a great medical need to actually improve cognitive functions in people that still suffer from persistent cognitive impairments one year after a stroke.

Animal studies have shown that the enzyme phosphodiesterase type 4 (PDE4) plays an important role in the brain, as it has been shown to be critically linked to neuronal plasticity. Although animal studies may not always predict effects in humans, there is a strong case that PDE4 inhibition may also work in humans. Researchers from Maastricht University, and others, have shown that the PDE4 inhibitor roflumilast improved memory performance in old healthy participants and in schizophrenic patients. This is a proof of concept that PDE4 inhibition can improve memory performance in humans. A logical next step is to test if roflumilast can improve cognitive functioning and daily life activities in people suffering from cognitive problems more than one year after stroke.

Objective: The objective is to validate the effects of chronic roflumilast treatment on cognitive function (i.e. episodic memory) by means of behavioral tasks, in people suffering from cognitive impairments at least 1 year after stroke. Secondary, the effects of roflumilast on daily activities and well-being will be assessed.

Study design: The first phase of study will be conducted according to a double-blind, randomized placebo-controlled, between-subjects design. In a second phase, the placebo group will be given the opportunity to receive roflumilast. This is an open label design.

Study population: 100 female and male, people (41-70 years old) suffering from cognitive complaints 1 year after stroke will be recruited via advertisements via social media and via local caretaking organizations (e.g., SGL, Adelante).

Intervention: The study will consist of 2 arms (N = 50 per arm): placebo and 100 μg roflumilast. The duration of treatment is planned for 3 months and participants will be tested at baseline, after 1.5 months, after 3 months. The participants will also do daily computer games to stimulate their brain function. The roflumilast group will be tested 3 months treatment stopped to test if the effects last after treatment is discontinued. After the end of the 3 months-intervention period, the participants of the placebo group will be identified and they will be asked whether they would like to take roflumilast for a 3-month period. This will give information as to the roflumilast effects in an open label setting. Moreover, this gives the participants in the placebo group the opportunity to receive the active treatment (if they wish)."

ELIGIBILITY:
Inclusion Criteria:

* Willingness to sign an informed consent
* Body mass index (BMI) between 18.5 and 35
* Suffered a stroke at least one year ago; and at the age of 40 or later
* Objective cognitive complaint: memory performance on the delayed recall in the 15 words VWLT of below the normative score (corrected for education, sex and age)

Exclusion Criteria:

* Normal Pressure Hydrocephalus (NPH)
* Morbus Huntington
* Parkinson's disease
* HIV/AIDS
* Hepatitis C & B
* Recent Transient Ischemic Attack (TIA) (< 1 years)
* Cerebrovascular Accident (<1 years)
* Chronic Obstructive Pulmonary Disease (COPD) type Gold 3 and 4
* History of schizophrenia, bipolar disorder or psychotic symptoms not otherwise specified or previous treatment for these diseases (lifetime)
* Risk of suicidal behaviour
* Current affective disorder (i.e. anxiety or major depression)
* Cognitive problems due to alcohol abuse, brain tumor, epilepsy, encephalitis or lack of capacity to consent to participation.
* Current treatment with (or illicit use of) cannabis, opiates, benzodiazepines, MDMA and cocaine
* Patients with moderate or major liver impairments will be excluded (e.g. Child-Pugh B and C).
* Use of medication showing strong inhibition of either CYP3A4 or CYP1A2
* Patients with rare hereditary problems of galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption
* Patients participating in other drug studies

Ages: 41 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-07-07 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Verbal Learning Test (VLT) Verbal Learning Test (VLT) (15 words) (delayed recall) [ Time Frame: Change from baseline to 12 weeks of chronic intake ] Verbal Learning Test (VLT) | Change from baseline to 12 weeks of chronic intake
  15 words, delayed recall

SECONDARY OUTCOMES:
Verbal Learning Test (VLT) | Change from baseline to effects one hour after the first intake (acute effects), to 6 weeks of chronic intake and to 12 weeks after the end of treatment (long-term effects)
  15 words, delayed recall
Rivermead Behavioural Memory Test | Change from baseline to effects one hour after the first intake (acute effects), to 6 weeks of chronic intake, to 12 weeks of chronic intake and to 12 weeks after the end of treatment (long-term effects)
Digit Symbol Substitution Test (DSST) | Change from baseline to effects one hour after the first intake (acute effects), to 6 weeks of chronic intake, to 12 weeks of chronic intake and to 12 weeks after the end of treatment (long-term effects)
Trail Making Test (TMT) | Change from baseline to effects one hour after the first intake (acute effects), to 6 weeks of chronic intake, to 12 weeks of chronic intake and to 12 weeks after the end of treatment (long-term effects)
Everyday Memory Questionnaire | Change from baseline to effects one hour after the first intake (acute effects), to 6 weeks of chronic intake, to 12 weeks of chronic intake and to 12 weeks after the end of treatment (long-term effects)
the total mood score of the Hospital Anxiety and Depression Scale questionnaire (HADS) | Change from baseline to effects one hour after the first intake (acute effects), to 6 weeks of chronic intake, to 12 weeks of chronic intake and to 12 weeks after the end of treatment (long-term effects)
Mood and well-being: Utrecht Scale for Evaluation of Rehabilitation-Participation (USER-Participation) (USER-P) | Change from baseline to effects one hour after the first intake (acute effects), to 6 weeks of chronic intake, to 12 weeks of chronic intake and to 12 weeks after the end of treatment (long-term effects)

CONTACTS AND LOCATIONS:
Overall Officials: Ieke Winkens, Dr., Principal Investigator — Assistant Professor
Locations (1):
- Maastricht University, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No